CLINICAL TRIAL: NCT04557904
Title: Effects of Craniocervical Flexion Exercises and Scapular Stabilization Exercises in Neck Pain and Forward Head Posture Among Female Wearing Head Scarves
Brief Title: Comparison of Craniocervical Flexion and Scapular Stabilization Exercises in Forward Head Posture and Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/18/1006 Sanjeela Abbas
Record Dates: First submitted 2020-09-16; First posted 2020-09-22 (Actual); Last update posted 2020-09-22 (Actual); Status verified 2020-09

CONDITIONS: Cervical Pain
Keywords: Forward head posture, Craniocervical flexion exercises
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: Craniocervical flexion exercises (Experimental): Exercise protocol were performed over a 4 week duration under the command of a supervisor. Subjects were asked not to obtain any other particular intervention for cervical ache. Command the subject to be in crook lying position. Lock their finger to place their finger below the skull and retract the lower jaw and retract chin as far as possible.
  Interventions: Other: Craniocervical flexion exercises
- Group B: Scapular stabilization exercises (Experimental): Group B performed scapular stabilization workout for 30 minutes per session, three days a week for four weeks. The scapular stabilization exercises were made up of four stages
  Interventions: Other: Scapular stabilization exercises

INTERVENTIONS:
Other: Craniocervical flexion exercises — Command the subject to be in crook lying position. Lock their finger to place their finger below the skull and retract the lower jaw and retract chin as far as possible. Subject has to slightly raise his/he skull a few centimeters. Fingers should be touching the cranium but not supporting it. Subject had to respire and hold the position. Subject has the move out the chin. Stop exercise and restart again. Perform this exercise for 10 times by holding this position for 20 sec at the start of the exercise, increasing it by 10 seconds every session commonly underwent pectoralis minor stretching before every session of exercise of 4 sets with 30 second's hold
  Arms: Group A: Craniocervical flexion exercises
Other: Scapular stabilization exercises — The scapular stabilization exercises were made up of four stages: (1) In supine position, the patient was commanded to deep respire for the sake of relaxation by maintain the cervical and shoulder in relaxing position to take a deep breath to relax the body while holding her shoulders and neck in relaxing position. (2) The patient then flex her knees and placed her feet flat on the plinth, and maintain the pose without any cervical movement. Then the patient asked to raise her dominant arm to 90° shoulder flexion with full elbow extension and scapular protraction. This position was sustained for 10 seconds before going to initial position. Three laps of 10 repetitions with one-minute interval in between were performed. (3) In quadruped position, the patient raise her arms alternatively with shoulder abduction and 120 ° flexion. That posture was held for 10 seconds before returning to the starting position. (4) In sitting position
  Arms: Group B: Scapular stabilization exercises

SUMMARY:
The aim of this research is to compare the effects of craniocervical flexion exercises and scapular stabilization exercises in reducing neck pain and forward head posture among females wearing head scarves. Quasi experimental trials done at Akhtar Saeed Trust hospital, Falah o Behbud Associations and Medicare Hospital (Lahore, Pakistan). A sample size of 50 patients was taken using non-probability purposive sampling technique. Subjects were randomly divided into 2 groups. Subjects in group A were treated with craniocervical flexion exercises and the subjects in group B were treated with scapular stabilization exercises with 25 subjects in each group. Pretreatment evaluation was done using numeric pain rating scale (NPRS) and neck disability index (NDI) as subjective measurement and Goniometry for assisted range of motion (AROM) and plumb line method for measuring head posture as objective measurement. The baseline values for all dependent variables were recorded on day one and at the end of 4th week.

DETAILED DESCRIPTION:
Neck pain is very common problem which is characterized by pain and soreness, felt in the area that lies between the lower margin of the occiput and 1st thoracic vertebra. Forward head posture can take place when head translated anteriorly and lower cervical spine goes into flexion or both and it is thought to be related with an increase in upper cervical spine extension. Most common abnormality which is associated with neck pain is forward head posture also known as chin poking. In which head is protrude out in sagittal plane and placed anteriorly to the trunk. It is considered that forward head posture causes an increase in compressive forces on the apophyseal joints of cervical spine and also on the posterior portion of vertebra. That is why, the length and strength of connective tissue change (due to the stretching of anterior structures and shortening of posterior muscles of neck ) following the pain. Shoulder blades and thoracic spine may also be affected with forward head posture, generally causing the imbalance in musculoskeletal system. Cervical flexor and extensor muscle groups strength & endurance performance ratio determined the magnitude of forward head posture . During daily activities the prolonged static posture in neck , shoulders and head may cause neck pain. Neck pain persistence is often considered to be associated with abnormalities in head posture, therefore some clinicians emphasized its importance while during examination. Postural effects on health is becoming more apparent and the most frequent postural problem is forward neck posture, occurring in between 66-90% of the population approximately. However, with increasing age the cervical range of motion decreased and it's prevalence increased with longer disease period. Generally, the neck pain is more prevalent in women than men. Wearing the headscarf is a part of an essential religious practice by females in Islamic cultures. The headscarf is referred to the scarf that wraps up over the head and around the neck. According to the Pew Research Center there are approximately 1.7 billion Muslims in the world. Estimating the total number of females worldwide who wear headscarves is difficult. Several Islamic countries mandate females to wear headscarves when out in public, while other countries have banned the use of headscarves in public. However, in the majority of the world's countries, wearing headscarves is optional. Females in Islamic cultures wear the headscarf when they are in public and usually begin wearing it at the onset of puberty. Regular wear of the headscarf might have an influence on cervical proprioception and range of motion (ROM). Recent studies have identified impaired activation of the deep cervical flexor muscles, the longus colli and longus capitis, in people with neck pain. Craniocervical flexion is the principal action of deep cervical muscles. Given the role of the deep cervical flexor muscles in postural support and the knowledge of impaired activation of these muscles in people with neck pain, it is likely that this patient population also would display deficits in the postural endurance of these muscles and painful cervical spine disorders. Indeed, evidence suggests that people with neck pain drift into a more forward head position when distracted and Craniocervical flexion exercises improves forward head posture and reduce neck pain.Moreover, retraining the deep cervical flexor muscles, which has been shown to decrease neck symptoms and increase the activation of the deep cervical flexor muscles during performance of the clinical test of craniocervical flexion, may improve the ability to maintain an upright posture of the cervical spine. Furthermore, there is a relationship between cervical ROM and forward head posture.Repeated upper cervical retractions (strengthening deep cervical flexors and stretching cervical extensors) changed resting neck posture. Scapular stabilization brought about improvement in posture through activation of the neck muscles, the lower trapezius, and the serratus anterior. Therefore, this intervention has a positive effect on neck alignment by reducing the compensatory movements of the muscles involved in forward head posture. There is a lack of literature regarding neck pain and forward head posture in females wearing head scarves . That is why, in this study,Forward head posture measurements will be obtained. In addition, the effect of interventions to improve cervical muscle flexibility in this population will be explained. In this study, we considered three factors related to headscarves, Onset of the practice, hours worn per day, and the number of years worn.

LITERATURE REVIEW

In 2017 determined the effects of wearing the headscarf on cervical spine ROM and joint position error. To analyze the influence of age at onset of wearing the headscarf and duration of hours per day wearing the headscarf on cervical range of motion and joint position error. The headscarf group reported a significant limitation in cervical range of motion in all six directions. Joint position error test revealed no significant difference between groups. Moreover, females in the headscarf group who wore the headscarf for more than 6 hours per day had significantly less left rotation compared to those who wear it for less than or equal to 6 hours, Wearing of the headscarf may result in cervical range of motion limitation. The duration of wearing the headscarf daily is a key factor to limited cervical range of motion an increase in cervical Joint position error.

In 2017 determined the effect of forward head posture-improving exercises on rounded shoulder posture when employing the self-stretch exercise, the McKenzie exercise, and the Kendall exercise as intervention methods based on previous studies that reported negative effects of unbalanced posture and musculoskeletal problems on forward head posture and rounded shoulder posture. Their study results showed that all interventions increased the craniovertebral angle and the scapular index, which revealed that the applied exercises had a positive effect on forward head posture and rounded shoulder posture.

In 2018, designed the basic data for developing exercise program that helps correcting posture by knowing the effect of strengthening and elongation exercises of upper extremity muscle to forward head posture correction. After 4 weeks of neck and chest extensor muscle exercise, the group who exercised both showed increase in range of neck joint motion and neck flexion of the forward head posture. However, this study provides the fact that the group who exercised both neck and chest muscle had more effect than the control group.

In 2017 evaluated the effects of a 16-week resistance and stretching training program applied in physical education (PE) classes on forward head posture and protracted shoulder posture in Portuguese adolescents.. Study concluded that A 16-week resistance and stretching training program decreased forward head and protracted shoulder postures in adolescents.

In 2017 , evaluated the effect of modified cervical exercise and determine whether such exercise improves the range of motion of the cervical movement in smartphone users with forward head posture.According to the results of this study,A significantly increased range of motion was seen in all three groups that performed the modified cervical exercises, although the modified cervical exercises were performed for only a relatively short duration (four weeks), the exercises brought about an improvement in the forward head posture that was induced by using a smartphone.

In 2018 investigated the effects of scapular stabilization exercise on neck posture, muscle activity, pain, and quality of life in individuals with neck pain and forward head posture. Training the scapular stabilization group showed significant improvement on the craniovertebral angle, upper trapezius muscle activity, serratus anterior muscle. Study concluded that Scapular stabilization exercise can help improve the head posture and pain in the patients with neck pain and forward head posture. Controlling the muscular activities through scapular stabilization exercise also improves the patients' quality of life.

In 2018 investigated the effects of scapula movement on neck alignment and the muscles in patients with forward head posture, who has the structural changes around the neck caused from the forward head posture, when scapular stabilization exercise is applied. Scapular stabilization brought about improvement in posture through activation of the neck muscles, the lower trapezius, and the serratus anterior. Therefore, the intervention has a positive effect on neck alignment by reducing the compensatory movements of the muscles involved in forward head posture.

ELIGIBILITY:
Inclusion Criteria:

* Forward-head-posture
* Duration of wearing-the headscarf/hijab for a minimum of 5-years
* Females ho start wearing headscarf before or at the age of-20. Females having neck-pain for less-than-six-months or if they had any muscular spasm & tenderness in the neck region.
* Pain being experienced in cervical spine area, which started from-superior-nuchal line-to the first thoracic vertebra.
* Pain radiating with or without any extensive radicular-symptoms towards other areas of body such as head and upper extremities.
* Restricted range-of-motion of cervical-spine.

Exclusion Criteria:

* Any red flags (tumor, osteoporosis, metabolic disorders, fracture, rheumatoid arthritis, resting-blood-pressure higher than 140/90 mmHg, prolonged-history of steroids abuse, continuous nerve root entrapment with two-or more-positive-neurologic-signs (muscle weakness involving cervical myotomes, abnormal upper limb deep-tendon-reflexes, or- -abnormal cervical dermatome.
* Already diagnosed with cervical spine-stenosis, showed bilateral upper limb symptoms.
* Any six weeks prior history of whiplash-injury or engaged in any type of treatment regarding neck pain from any-practitioner within the last month.
* History-of any previous-cervical or thoracic-spine-surgery-

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2018-06-15 (Actual); Primary Completion 2019-02-20 (Actual); Study Completion 2019-03-15 (Actual)

PRIMARY OUTCOMES:
Neck disability index | 4th week
  Changes from base line Northwick disability index was developed first in Northwick Park hospital, England. It was designed to measure the neck pain and disability over time. It consists of 10, five parts sections. At the end, score is calculated by dividing the obtained score by total (50) multiplied by 100. As the driving section was missing in all the female patients, total score was considered as 45 instead of 50
Numeric Pain Rating Scale | 4th week
  Changes from base Line Numeric Pain rating scale is a scale for pain starting from 0-10. where 0 indicate no pain and 10 indicate severe pain.
ROM Cervical Spine ( Flexion) | 4th week
  Changes from the Baseline ROM range of Motion of Cervical spine flexion was taken with the Help of Goniometer
ROM Cervical Spine ( extension) | 4th week
  Changes from the Baseline ROM range of Motion of Cervical spine extension was taken with the Help of Goniometer
ROM Cervical Spine ( Right side flexion) | 4th week
  Changes from the Baseline ROM range of Motion of Cervical spine right side flexion was taken with the Help of Goniometer
ROM Cervical Spine ( left side Flexion) | 4th week
  Changes from the Baseline ROM range of Motion of Cervical spine left side flexion was taken with the Help of Goniometer
ROM Cervical Spine ( right rotation) | 4th week
  Changes from the Baseline ROM range of Motion of Cervical spine right rotation was taken with the Help of Goniometer
ROM Cervical Spine ( left rotation) | 4th week
  Changes from the Baseline ROM range of Motion of Cervical spine left rotation was taken with the Help of Goniometer
Plumb Line | 4th week
  Participants were requested to wear the suitable attire to properly expose the areas being examined e.g thoracic & cervical spine. The lobe of ear, the seventh cervical vertebra, acromion process, the thoracic spine and lateral malleolus were used as landmarks for measuring the head posture

CONTACTS AND LOCATIONS:
Overall Officials: Rabiya Noor, PHD, Principal Investigator — Riphah International University
Locations (1):
- Akhtar Saeed Trust hospital, Falah o Behbud Associations and Medicare Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nejati P, Lotfian S, Moezy A, Moezy A, Nejati M. The relationship of forward head posture and rounded shoulders with neck pain in Iranian office workers. Med J Islam Repub Iran. 2014 May 3;28:26. eCollection 2014. PMID 25250268
- [Background] Kim JY, Kwag KI. Clinical effects of deep cervical flexor muscle activation in patients with chronic neck pain. J Phys Ther Sci. 2016 Jan;28(1):269-73. doi: 10.1589/jpts.28.269. Epub 2016 Jan 30. PMID 26957772
- [Background] Lopez-de-Uralde-Villanueva I, Beltran-Alacreu H, Paris-Alemany A, Angulo-Diaz-Parreno S, La Touche R. Relationships between craniocervical posture and pain-related disability in patients with cervico-craniofacial pain. J Pain Res. 2015 Jul 30;8:449-58. doi: 10.2147/JPR.S84668. eCollection 2015. PMID 26261425
- [Background] Dunleavy K, Goldberg A. Comparison of cervical range of motion in two seated postural conditions in adults 50 or older with cervical pain. J Man Manip Ther. 2013 Feb;21(1):33-9. doi: 10.1179/2042618612Y.0000000017. PMID 24421611
- [Background] Benatto MT, Florencio LL, Bragatto MM, Dach F, Fernandez-de-Las-Penas C, Bevilaqua-Grossi D. Neck-specific strengthening exercise compared with sham ultrasound when added to home-stretching exercise in patients with migraine: study protocol of a two-armed, parallel-groups randomized controlled trial. Chiropr Man Therap. 2020 May 19;28(1):22. doi: 10.1186/s12998-020-00313-w. PMID 32423454
- [Background] Blomgren J, Strandell E, Jull G, Vikman I, Roijezon U. Effects of deep cervical flexor training on impaired physiological functions associated with chronic neck pain: a systematic review. BMC Musculoskelet Disord. 2018 Nov 28;19(1):415. doi: 10.1186/s12891-018-2324-z. PMID 30486819
- [Background] Suvarnnato T, Puntumetakul R, Uthaikhup S, Boucaut R. Effect of specific deep cervical muscle exercises on functional disability, pain intensity, craniovertebral angle, and neck-muscle strength in chronic mechanical neck pain: a randomized controlled trial. J Pain Res. 2019 Mar 7;12:915-925. doi: 10.2147/JPR.S190125. eCollection 2019. PMID 30881101
- [Background] Rudolfsson T, Bjorklund M, Svedmark A, Srinivasan D, Djupsjobacka M. Direction-Specific Impairments in Cervical Range of Motion in Women with Chronic Neck Pain: Influence of Head Posture and Gravitationally Induced Torque. PLoS One. 2017 Jan 18;12(1):e0170274. doi: 10.1371/journal.pone.0170274. eCollection 2017. PMID 28099504
- [Background] Yang CC, Su FC, Yang PC, Lin HT, Guo LY. Characteristics of the Motor Units during Sternocleidomastoid Isometric Flexion among Patients with Mechanical Neck Disorder and Asymptomatic Individuals. PLoS One. 2016 Dec 12;11(12):e0167737. doi: 10.1371/journal.pone.0167737. eCollection 2016. PMID 27941995
- [Background] Hidalgo B, Hall T, Bossert J, Dugeny A, Cagnie B, Pitance L. The efficacy of manual therapy and exercise for treating non-specific neck pain: A systematic review. J Back Musculoskelet Rehabil. 2017 Nov 6;30(6):1149-1169. doi: 10.3233/BMR-169615. PMID 28826164
- [Background] Coulter ID, Crawford C, Vernon H, Hurwitz EL, Khorsan R, Booth MS, Herman PM. Manipulation and Mobilization for Treating Chronic Nonspecific Neck Pain: A Systematic Review and Meta-Analysis for an Appropriateness Panel. Pain Physician. 2019 Mar;22(2):E55-E70. PMID 30921975
- [Background] Groeneweg R, van Assen L, Kropman H, Leopold H, Mulder J, Smits-Engelsman BCM, Ostelo RWJG, Oostendorp RAB, van Tulder MW. Manual therapy compared with physical therapy in patients with non-specific neck pain: a randomized controlled trial. Chiropr Man Therap. 2017 Apr 28;25:12. doi: 10.1186/s12998-017-0141-3. eCollection 2017. PMID 28465824
- [Background] Groeneweg R, Kropman H, Leopold H, van Assen L, Mulder J, van Tulder MW, Oostendorp RA. The effectiveness and cost-evaluation of manual therapy and physical therapy in patients with sub-acute and chronic non specific neck pain. Rationale and design of a Randomized Controlled Trial (RCT). BMC Musculoskelet Disord. 2010 Jan 24;11:14. doi: 10.1186/1471-2474-11-14. PMID 20096136
- [Background] Price J, Rushton A, Tyros I, Tyros V, Heneghan NR. Effectiveness and optimal dosage of exercise training for chronic non-specific neck pain: A systematic review with a narrative synthesis. PLoS One. 2020 Jun 10;15(6):e0234511. doi: 10.1371/journal.pone.0234511. eCollection 2020. PMID 32520970
- [Background] Damgaard P, Bartels EM, Ris I, Christensen R, Juul-Kristensen B. Evidence of Physiotherapy Interventions for Patients with Chronic Neck Pain: A Systematic Review of Randomised Controlled Trials. ISRN Pain. 2013 Apr 15;2013:567175. doi: 10.1155/2013/567175. eCollection 2013. PMID 27335877
- [Background] Bernal-Utrera C, Gonzalez-Gerez JJ, Anarte-Lazo E, Rodriguez-Blanco C. Manual therapy versus therapeutic exercise in non-specific chronic neck pain: a randomized controlled trial. Trials. 2020 Jul 28;21(1):682. doi: 10.1186/s13063-020-04610-w. PMID 32723399